CLINICAL TRIAL: NCT02704052
Title: Real-time Anti-Factor Xa Measurements in Surgical Patients to Examine Enoxaparin Metabolism and Optimize Enoxaparin Dose
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Pannucci, M.D., University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00086103
Record Dates: First submitted 2016-03-07; First posted 2016-03-09 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Deep Venous Thrombosis; Pulmonary Embolus; Venous Thromboembolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard enoxaparin dose (Active Comparator): We will identify a convenience sample of surgical patients placed on enoxaparin prophylaxis at their attending surgeon's discretion-the proposed research will not dictate the initial enoxaparin dose magnitude or frequency. However, we will identify patients already on enoxaparin, evaluate peak and trough steady state aFXa levels, and adjust patient's dose if necessary based on steady state aFXa levels. Eligible patients will have enoxaparin prophylaxis started within 36 after surgery at their surgeon's discretion. Steady state peak and trough aFXa levels will be drawn at 4 and 12 hours, respectively, after the third enoxaparin dose. Goal peak aFXa levels will be 0.2-0.4 IU/mL for twice daily dosing and 0.3-0.5 IU/mL for once daily dosing.
  Interventions: Drug: Standard enoxaparin dose
- Real time enoxaparin dose adjustment (Experimental): Patients with identified out of range levels will receive pharmacist-driven real time enoxaparin dose adjustment and will receive followup steady state peak and trough aFXa levels. aFXa monitoring will be discontinued when in range peak levels are obtained, when enoxaparin prophylaxis is discontinued at surgeon discretion, or when the patient is discharged. Patients may be continued on enoxaparin prophylaxis after discharge per attending surgeon discretion but aFXa levels will not be followed in the outpatient environment.
  Interventions: Drug: Real time enoxaparin dose adjustment

INTERVENTIONS:
Drug: Real time enoxaparin dose adjustment — Patients will have steady state peak and trough anti-Xa levels drawn after their third enoxaparin dose. Patients with out of range peak anti-Xa levels will receive real time enoxaparin dose adjustment followed by repeat peak and trough anti-Xa levels.
  Arms: Real time enoxaparin dose adjustment
Drug: Standard enoxaparin dose — Patients will be placed on enoxaparin prophylaxis per their surgeon's discretion.
  Arms: Standard enoxaparin dose

SUMMARY:
Venous thromboembolism (VTE) encompasses deep venous thrombosis and pulmonary embolus, and is the proximate cause of death in over 100,000 hospitalized patients per year.

This project will critically examine the pharmacokinetics of prophylactic doses of enoxaparin in surgical patients, and will evaluate how alteration of enoxaparin dose magnitude and frequency affects peak and trough aFXa levels as well as risk for re-operative hematoma. If subtherapeutic aFXa levels are observed, the study will design, implement and test a clinical protocol to optimize post-operative aFXa levels. Although not an explicit Aim, this study will also provide important preliminary data on VTE rates in surgical patients with in range and out of range aFXa levels.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) encompasses deep venous thrombosis and pulmonary embolus, and is the proximate cause of death in over 100,000 hospitalized patients per year. To put this in better context, VTE kills more people each year than the annual morbidity from motor vehicle crashes and breast cancer combined. Surgeons commonly provide enoxaparin, a low molecular weight heparin, for VTE prophylaxis. Enoxaparin's activity is quantified by anti-Factor Xa (aFXa) levels. Studies of enoxaparin metabolism in patients with traumatic injury, thermal injury, or those undergoing reconstructive surgery have shown that standard dosing can result in inadequate aFXa levels, likely from the hypermetabolic state associated with significant injury. Small studies have associated subtherapeutic aFXa levels with increased risk for life or limb-threatening VTE events. Prior work from has shown that 2-10% of highest risk surgical patients have a VTE event despite enoxaparin prophylaxis. The investigators believe that surgical patients would benefit from an individualized dosing regimen for enoxaparin prophylaxis and that individualized dosing will decrease observed rates of life or limb-threatening post-operative VTE events.

This project will critically examine the pharmacokinetics of prophylactic doses of enoxaparin in surgical patients, and will evaluate how alteration of enoxaparin dose magnitude and frequency affects peak and trough aFXa levels as well as risk for re-operative hematoma. If subtherapeutic aFXa levels are observed, the study will design, implement and test a clinical protocol to optimize post-operative aFXa levels. Although not an explicit Aim, this study will also provide important preliminary data on VTE rates in surgical patients with in range and out of range aFXa levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults, (age≥18)
* Patients who have had surgery with general anesthesia.
* Post-operative stay will be ≥2 days

Exclusion Criteria:

* Contradiction to use enoxaparin
* History of intracranial bleeding/stroke, hematoma or bleeding disorder, heparin-induced thrombocytopenia positive, and heparin-induced thrombocytopenia positive
* Creatinine clearance ≤ 30mL/min
* Serum creatinine >1.6mg/dL
* Epidural anesthesia
* Patients placed on non-enoxaparin chemoprophylaxis regimens per their surgeon's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism | 90 days
  Symptomatic 90-day VTE confirmed with imaging

SECONDARY OUTCOMES:
Re-operative hematoma | 90 days
  Bleeding requiring return to the operating room within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Puccini, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospitals, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pannucci CJ, Fleming KI, Varghese TK Jr, Stringham J, Huang LC, Pickron TB, Prazak AM, Bertolaccini C, Momeni A. Low Anti-Factor Xa Level Predicts 90-Day Symptomatic Venous Thromboembolism in Surgical Patients Receiving Enoxaparin Prophylaxis: A Pooled Analysis of Eight Clinical Trials. Ann Surg. 2022 Dec 1;276(6):e682-e690. doi: 10.1097/SLA.0000000000004589. Epub 2020 Oct 19. PMID 33086312
- [Derived] Pannucci CJ, Fleming KI, Bertolaccini CB, Prazak AM, Huang LC, Pickron TB. Assessment of Anti-Factor Xa Levels of Patients Undergoing Colorectal Surgery Given Once-Daily Enoxaparin Prophylaxis: A Clinical Study Examining Enoxaparin Pharmacokinetics. JAMA Surg. 2019 Aug 1;154(8):697-704. doi: 10.1001/jamasurg.2019.1165. PMID 31116389